CLINICAL TRIAL: NCT06187428
Title: The PainSMART Project: A Research Program on Effectiveness, Mechanisms of Effect and Patient-practitioner Experiences of the PainSMART-strategy as an Adjunct to Usual Primary Care Physiotherapy Management for Musculoskeletal Pain
Brief Title: The PainSMART Research Program: Evaluating a Pain Education Strategy for Patients Seeking Primary Care Physiotherapy
Acronym: PainSMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kajsa Johansson (Other Government)
Collaborators: The Research Council of South East Sweden (FORSS) (Unknown)
Responsible Party: Sponsor-Investigator, Kajsa Johansson, Senior associate Professor, Linkoeping University
Organization: Linkoeping University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dnr 2023-05968-01; Primary care rehabilitation (Other: County council of Östergötland); Primary care rehabilitation (Other: County council of Jönköping)
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Pain; Pain Acute; Pain, Chronic; Self Efficacy; Illness Perceptions; Physical Activity Level; Sickness Absence; Referral and Consultation; Worry; Anxiety; Patient-Centered Care; Communication
Keywords: pain; education; pain self efficacy; digitalisation; primary care
MeSH Terms: conditions — Pain; Acute Pain; Chronic Pain; Anxiety Disorders; Communication

STUDY DESIGN:
Intervention Model Description: Two-arm parallel randomised assignment to intervention (PainSMART) group or control (usual management) group
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes are collected digitally and pseudonymised and the statistical analyses will be blinded to group allocation since the randomisation is concealed during this process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PainSMART-strategy (intervention) group (Experimental): Patients eligible for inclusion first contact the physiotherapy department and are triaged by a physiotherapist and booked for an initial physiotherapy consultation. After triage, study information and the consent to participate, patients randomised to the intervention group receive the PainSMART-strategy as an adjunct to usual MSKP physiotherapy management.
  The strategy includes; exposure to the film 'Be PainSMART:er' at baseline, together with ratings of the clarity of the film's key-messages, a second film exposure prior to the initial consultation and three questions related to the film at the initial consultation.
  Baseline data collection will occur prior to first exposure to the film. The film is available exclusively via the questionnaires via Region Östergötland's Quick channel. Therefore it is not shareable or available via online searching.
  Interventions: Other: PainSMART-strategy
- Usual physiotherapy management (control) group (Active Comparator): Patient participants randomised to the control group will follow the usual physiotherapy management pathway at the physiotherapy departments participating in the study.
  Interventions: Other: Usual physiotherapy management

INTERVENTIONS:
Other: PainSMART-strategy — Be PainSMART:er is a seven minute long film developed by the research group based on modern pain science and previous qualitative studies.
  The film is divided into three sections:
  Section 1- Educates that MSKP is a complex protective system that does not reflect the anatomical state of the body and provides reassurance that MSKP is rarely caused by serious pathology.
  Section 2- Provides advice on active MSKP coping, such as encouraging work despite some pain, in an attempt to reconceptualise the belief that a painful body part needs to be rested.
  Section 3- Aims to prepare patients for a biopsychosocial physiotherapy consultation by encouraging them to reflect on the film's messages.
  In addition to the film, the questions posed to the participant at the initial consultation aim to facilitate the discussion around the film and MSKP reflections. Management subsequent to the initial consultation will follow usual management.
  Arms: PainSMART-strategy (intervention) group
Other: Usual physiotherapy management — Patients randomised to the control group follow usual MSKP physiotherapy management. Specifically, patients first contact their physiotherapy department online or via telephone and are triaged by a certified physiotherapist and are booked for an initial physiotherapy consultation. After triage, study information and the consent to participate, patients in the control group receive online data collection questionnaires identical to those of the intervention group at baseline and prior to the consultation, excluding the film and the questions linked to the film. The initial consultation will take place as usual according to the preferences of the physiotherapist. The physiotherapist will pose one question at start of the consultation to acknowledge the completion of control group questionnaires. Management subsequent to the initial consultation will follow usual management.
  Arms: Usual physiotherapy management (control) group

SUMMARY:
The goal of this clinical trial is to test the PainSMART-strategy in a population of patients seeking primary care physiotherapy for pain related to muscles, joints and bones, so called musculoskeletal pain. The PainSMART-strategy consists of a digital educational film (entitled Be PainSMART:er) and a discussion based on the film at the initial physiotherapy consultation.

The main questions this clinical trial aims to answer are:

1. Can the PainSMART-strategy update knowledge and beliefs about pain and aid early stage self-management of pain for participants seeking primary care physiotherapy with benign musculoskeletal pain?
2. Can the PainSMART-strategy improve evaluations of the initial physiotherapy consultation for both the patient and physiotherapist?

Participating patients will be randomised into two groups. One group (intervention group) will receive the PainSMART-strategy as an adjunct to the current physiotherapy care pathway for musculoskeletal pain. The other group (control group) will follow the current physiotherapy care pathway. The two groups will be followed and compared over three months. Self-report questionnaires and data from central healthcare registers will be collected during and after the three-month period to analyse what effects the PainSMART-strategy can have on the following health outcomes:

* Pain levels
* Beliefs that one can remain active despite pain
* Knowledge about pain
* Worry about the seriousness of the pain
* Expectations regarding recovery
* Use of pain self-management strategies
* Levels of physical activity
* Absence from work due to pain
* Number of referrals made for scans or x-rays, or to a specialist, for pain
* Number of healthcare visits and direct costs incurred for pain during the trial period.

Participating patients (both groups) and physiotherapists will also complete questionnaires to evaluate the effect of the PainSMART-strategy on the initial physiotherapy consultation.

The final 30 to 40 participating patients in the study will also have their initial consultation with the physiotherapist audio recorded in order to enable analysis of any potential influence of the PainSMART-strategy on communication around pain during the consultation.

DETAILED DESCRIPTION:
For more detailed information about the study see the attached study protocol and the attached statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* Patients who, via telephone or online text-based triage, are judged to have benign MSKP and are booked for an initial physiotherapy consultation at one of the five participating physiotherapy departments
* Adult patients (18 years or older)

Exclusion Criteria:

* Patients who are judged to require urgent medical examination due to suspected serious pathology (red flags)
* Patients who are booked to an initial physiotherapy consultation on the same day as, or the day directly following triage.
* Patients referred for physiotherapy following consultation with a tertiary care practitioner (e.g. orthopaedic surgeon, rheumatologist, neurologist)
* Patients who cannot communicate in Swedish to the equivalent of a 12-year-old native speaker (as judged by the triaging physiotherapist)
* Patients who, through visual impairments, are unable to complete the necessary questionnaires for the study
* Patients who are booked for an initial consultation with a physiotherapist who has not consented to taking part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline and proportion of responders in self-reported Pain Self-efficacy measured using the Pain Self-efficacy questionnaire 10 (PSEQ-10) (within- and between group changes) | The PSEQ-10 will be collected at baseline, 24-72 hours prior to the initial physiotherapy consultation, 24 hours post-initial physiotherapy consultation and again at three months post-baseline
  Pain self-efficacy will be measured using the PSEQ-10 (Nicholas, 2007). The PSEQ-10 is a self-reported ten item scale scored as a total (0-60) with a higher score indicating greater pain self-efficacy (higher score = better outcome). The PSEQ-10 includes ten statements where patients are asked to rate, from zero to six, how confident they are that they can do certain things despite their pain.
  Change = Baseline score compared to score 24-72 hours prior to the initial physiotherapy consultation, 24 hours post-initial physiotherapy consultation (primary outcome point 1) and again at three months post-baseline (primary outcome point 2).
  Secondary analyses of within and between-group differences in proportion of responders will be conducted based on the study specific minimal clinical important difference (MCID) for primary outcomes at primary outcome time points. The MCID will be calculated for the whole cohort using an anchor method based on Global rating of change scores.
Mean change from baseline and proportion of responders in self-reported Pain Intensity measured using numerical rating scale (NRS) (within- and between group changes) | NRS will be collected at baseline, 24-72 hours prior to the initial physiotherapy consultation, 24 hours post-initial physiotherapy consultation and again at three months post-baseline
  Self-reported average pain intensity (primary outcome), worst pain intensity and best pain intensity in the previous 24 hours will be measured using three separate Numerical Rating Scales (NRS) (0-10; 0 = no pain to 10 = worst imaginable pain). NRS rating related to the past 24 hours has been chosen to avoid overlap of the ratings at the separate data collection time points.
  Change = Baseline score compared to score 24-72 hours prior to the initial physiotherapy consultation, 24 hours post-initial physiotherapy consultation (primary outcome point 1) and again at three months post-baseline (primary outcome point 2).
  Secondary analyses of within and between-group differences in proportion of responders will be conducted based on the study specific minimal clinical important difference (MCID) for primary outcomes at primary outcome time points. The MCID will be calculated for the whole cohort using an anchor method based on Global rating of change scores.

SECONDARY OUTCOMES:
Mean change from baseline in self-reported Musculoskeletal pain illness perceptions measured using the Brief Illness Perception Questionnaire (BIPQ) (within- and between group changes) | BIPQ will be collected at baseline, repeated directly after first exposure to the film, 24-72 hours prior to the initial physiotherapy consultation, 24 hours post-initial physiotherapy consultation and again at three months post-baseline
  The BIPQ has nine questions, eight use an 11-point NRS with anchor statements. Question 9 is a free text question where participants list the three most important factors they believed cause their MSKP (Broadbent et al., 2006).
  Change = Baseline score compared to score 24-72 hours prior to the initial physiotherapy consultation, 24 hours post-initial consultation and again at three months post-baseline.
  BIPQ will be analysed as recommended by Broadbent et al (2015): As individual items and as total score (max 80). The total score gives an impression of the patient's perception of the threat level of their MSKP, with a higher score reflecting a higher threat (lower item or total score=better outcome). The causal item question will be collected at baseline, immediately following the baseline exposure to the film and again at 24 hours post-initial consultation. The causal item question will be analysed by grouping of answers into categories.
Mean change from baseline in self-reported level of reassurance as to the benign nature of MSKP will be measured using a single numerical rating scale (Reassurance NRS) (within- and between group changes) | Reassurance NRS will be collected at baseline, 24-72 hours prior to the initial physiotherapy consultation, 24 hours post-initial physiotherapy consultation and again at three months post-baseline.
  Self-reported level of reassurance about the seriousness of MSKP will be measured using a reassurance NRS with an eleven-point scale (0-10). The reassurance NRS asks the participant how certain they are that there is not a serious condition causing their MSKP. A higher score indicates greater assurance. This question has been adapted from the original research by Sox et al. (1981) and has been previously used in research on acute LBP (Deyo et al., 1987).
  Change =Baseline score compared to score 24-72 hours prior to the initial physiotherapy consultation, 24 hours post-initial physiotherapy consultation and again at three months post-baseline.
Mean change from baseline in self-reported traditional musculoskeletal pain coping strategies and psychological flexibility measured using the Brief Pain Coping Inventory 2 (BPCI-2) (within- and between group changes) | BPCI-2 will be collected at baseline, 24-72 hours prior to the initial physiotherapy consultation, 24 hours post-initial physiotherapy consultation and again at three months post-baseline.
  The BPCI-2 is a 19-item questionnaire, where participants are asked to report on how many days in the last week they adopted certain pain management strategies (0-7 days; Vowles et al., 2014). The BPCI-2 is scored as a total score (0-133) and also contains two sub-scales which measure traditional pain coping strategies (max 56) and psychological flexibility (max 77; with 4 reverse scored items). Higher total or sub-scale scores indicate more adaptive coping (Vowles et al., 2014).
  Change = Baseline score compared to score 24-72 hours prior to the initial physiotherapy consultation, 24 hours post-initial physiotherapy consultation and again at three months post-baseline.
Mean change in self-reported levels of physical activity measured using three screening questions developed for the Swedish national board of health and welfare (within- and between group changes) | Physical activity will be collected at baseline, 24-72 hours prior to the initial physiotherapy consultation, 24 hours post-initial physiotherapy consultation and again at three months post-baseline.
  The three questions ask the participants how many minutes in the last week they have performed activity that makes the breathless, how many minutes they have been otherwise physically active, for example house work or gardening, and how many hours they usually sit during a day (not including sleeping) (Kallings, 2014).
  Change = Within and between group mean change in the scores over time from baseline to follow-up three months post-baseline (all time points). Scores on question regarding "Moderate to intensive exercise" and "Other physical activity beside exercise" will also be converted to activity minutes per week < 150min/w or ≥ 150min/w.
Mean self-reported global rating of change measured using a global rating of change scale (GRoCs) measured at three time points (analysed for both within- and between group changes) | GRoCs will be collected at three time points; first 24-72 hours prior to the initial physiotherapy consultation, 24 hours post-initial physiotherapy consultation and again at three months post-baseline
  Global Rating of Change will be measured using a single item GRoCs scored on an 11-point scale. The 11-point scale is scored from minus five to plus five, anchored by the terms very much worse (minus five), unchanged (zero) and completely recovered (plus five) in accordance with the recommendation made by Kamper et al. (2009). The score is based on the time period from when the participant first contacted their physiotherapy department and were triaged to 24-48 hours prior to the initial physiotherapy consultation and again at three months post-baseline.
  The score will be dichotomized into improved (1-5) and unchanged/worse (-5-0).
Change in type and frequency of self-reported analgesic medication use (within and between group changes) | will be collected at baseline, 24-72 hours prior to the initial physiotherapy consultation, 24 hours post-initial physiotherapy consultation and again at three months post-baseline.
  Self-reported analgesic medication use (type and consumption) for the presenting MSKP complaint will be collected via two questions. The first question establishes analgesic consumption and consumption frequency quantified via one question with response options: Yes, on a regular basis; Yes, sometimes; or No. The type of analgesics taken for MSKP is established via one question with six response options: 1. Paracetamol, 2. NSAID, 3. Opioids, 4. Gabapentinoids/Tricyclic antidepressants/Serotonin-norepinephrine reuptake inhibitors 5. Don't know 6. Other.
  Change = Baseline consumption (type & regularity) compared to score 24-72 hours prior to the initial physiotherapy consultation, 24 hours post-initial physiotherapy consultation and again at three months post-baseline. Analgesic type will be grouped into 3 groups for analysis:
  1. Paracetamol, 2. NSAID, 3. Opioids/gabapentinoids/Tricyclic antidepressants/Serotonin-norepinephrine reuptake inhibitors.
Total days of Sickness absence for each group (intervention and control) from baseline to three months post-baseline (between group difference) | Total aggregated days (for all participants in each group) from baseline to three months post-baseline
  Data on sickness certification will be collected for each participating patient via the Swedish social security database (Försäkringskassan) following completion of patient and physiotherapist outcome measure data collection. In addition the participants will self-rapport if they are currently on sick leave for their presenting MSKP complaint at the time of baseline data collection, 24-72 hours prior to the initial physiotherapy consultation, 24 hours post-initial physiotherapy consultation and again at the three month post-baseline data collection.
Total number of referrals for diagnostic imaging for each group (intervention and control) from baseline to three months post-baseline (between group differences) | Total aggregated referrals (for all participants in each group) made between baseline and three months post-baseline
  Data will be collected for each participating patient via regional healthcare databases (Rebus Vård, Region Östergötland & Region Jönköpings län) following completion of patient and physiotherapist outcome measure data collection. The number of referrals made for diagnostic imaging for musculoskeletal diagnoses for each participant made during the time that elapses between baseline and three months post-baseline will be collected.
Total number of referrals to tertiary/specialist care for musculoskeletal pain for each group (intervention and control) from baseline to three months post-baseline (between group differences) | Total aggregated referrals (for all participants in each group) made between baseline and three months post-baseline
  Data will be collected for each participating patient via regional healthcare databases (Rebus Vård, Region Östergötland & Region Jönköpings län) following completion of patient and physiotherapist outcome measure data collection. The number of referrals made to tertiary/specialist care for musculoskeletal diagnoses for each participant made during the time that elapses between baseline and three months post-baseline will be collected.
Total number of healthcare consultations attended for musculoskeletal pain for each group (intervention and control) from baseline to three months post-baseline (between group differences) | Total aggregated healthcare consultations attended (for all participants in each group) between baseline and three months post-baseline
  Data will be collected for each participating patient via regional healthcare databases (Rebus Vård, Region Östergötland & Region Jönköpings län) following completion of patient and physiotherapy outcome measure data collection. The number of healthcare appointments attended for musculoskeletal diagnoses for each participant during the time that elapses between baseline and three months post-baseline will be collected. Patients will also self-report if they have attended healthcare consultations for their MSKP presenting complaint with healthcare practitioners who are not the physiotherapist involved in the trial.
Direct healthcare costs per patient | Total aggregated direct healthcare costs (for all participants in each group) between baseline and three months post-baseline
  Direct costs per patient for healthcare during the MSKP study period will be collected from the central healthcare database. A comparison will be made between the intervention and control groups to establish if the PainSMART-strategy can improve health outcomes and the effectiveness of the physiotherapy management pathway.
One-off screening at baseline with the Örebro Musculoskeletal pain screening questionnaire | Baseline only
  The Örebro Musculoskeletal pain screening questionnaire (ÖMPSQ) is a ten item questionnaire which assesses five constructs; self-perceived function, pain experience, distress, fear-avoidance beliefs and return to work expectancy (Linton et al., 2011). The ÖMPSQ was developed in a primary care setting and the questionnaire is scored from 0-100 where a higher score indicates higher risk for future work related disability (Linton et al., 2011).

OTHER OUTCOMES:
One-off Patient reported evaluation of the initial physiotherapy consultation | 24 hours post-initial physiotherapy consultation
  The patients (intervention and control groups) will evaluate the initial consultation via seven questions adapted and modified from the National Patient Survey, Sweden. The seven questions evaluate if the patients felt that they had the possibility to talk sufficiently about their MSKP, whether they felt included in decision making around their care, whether they had the opportunity to discuss any worries and concerns they had regarding their MSKP and to what extent they discussed what they themselves could do to improve their MSKP and health. The participants will also be asked if they felt they could reach a consensus in understanding with the physiotherapist regarding their MSKP, whether the physiotherapist considered their personal MSKP experiences and explained MSKP in a way that they could understand. The questions are answered on a scale of 0-10 with zero representing less positive evaluation and ten a fully positive evaluation in relation to each question.
One-off Physiotherapist reported evaluation of the initial physiotherapy consultation | 24 hours post-initial physiotherapy consultation
  The physiotherapist participants will evaluate the initial physiotherapy consultation via three questions adapted and modified from the National Patient Survey, Sweden.
  The physiotherapists will answer three questions rating whether they felt they received sufficient information from the patient to adequately make clinical judgements regarding the patient's MSKP, whether they and the patient could reach a consensus in understanding regarding the patients MSKP and whether they felt the patient actively took part in decision making regarding their care.
  The questions are answered on a scale of 0-10 with zero representing less positive evaluation and ten a fully positive evaluation in relation to each question.
Intervention's groups rating of the clarity of the film's key-messages | After the first exposure to the film at baseline for patient participants in the intervention group only
  The intervention group will answer eight questions where they rate the clarity of the film's key messages. The film's key-messages reflect the following domains from the common-sense model of self-regulation; MSKP Identity, Timeline, Consequences, Causes, Control and Emotional representations.
Qualitative exploration of the influence of the PainSMART-strategy on the initial physiotherapy consultation (final 30 to 40 patient participants only) | Audio recording during the initial physioterapy consultation for the final 30 to 40 patient participants in the RCT
  Naturally occurring audio recordings of the initial physiotherapy consultations will be collected using Dictaphones for the final 30 to 40 patient participants in the trial only. This data will be used to conduct qualitative exploration of if or how exposure to the PainSMART-strategy influences communication around pain at the initial physiotherapy consultation
One-off Physiotherapist reported evaluation of patients preparedness for the initial physiotherapy consultation | Collected after each physiotherapist has conducted their final PainSMART study consultation
  Physiotherapists' experiences of their perception of the participating patients' preparedness for the initial consultation will be collected via one question for the intervention group and one question for the control group. The question will ask the physiotherapists to rate, on a scale from zero to ten, to what extent they felt that the patients in the film respective control groups were prepared for their initial physiotherapy consultation. Specifically the question askes to what extent the patient seemed to have reflected over biopsychosocial factors that may have influenced their pain experience and its impact on function and wellbeing prior to the initial consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Kajsa Johansson, PhD, Study Chair — Linkoeping University; Richard M Thompson, MSc, Principal Investigator — Linkoeping University; Maria Fors, PhD, Principal Investigator — Linkoeping University; Allan Abbott, PhD, Study Director — Linkoeping University; Ann-Sofi Kammerlind, PhD, Study Director — Linkoeping University; Pia Tingström, PhD, Study Director — Linkoeping University
Locations (6):
- Sweden (6):
  - Bra Liv VC Tranås, Primary Care Physiotherapy department, Svärtinge, Jönköping County
  - Rehab Finspång, Primary Care Physiotherapy department, Finspång, Östergötland County
  - Rörelse och Hälsa, Primary Care Physiotherapy department, Linköping, Östergötland County
  - Linköping University, Linköping, Östergötland County
  - Rehab Väst, Primary Care Physiotherapy department, Motala, Östergötland County
  - Rehab Öst, Primary Care Physiotherapy department, Norrköping, Östergötland County

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be shared pseudonymised upon reasonable request after study completion and after finalising relevant research program publications. This will include background data, patient reported outcome measure data and patient and physiotherapist experience measure data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol has been uploaded in conjunction with submission of this registration and prior to the start of patient recruitment to the first phase on the RCT (January 19, 2024).
  An update to the study protocol has been uploaded prior to the start of patient recruitment to the qualitative phase of the RCT (September 25, 2024)
  A statistical analysis plan has been uploaded to Clinicaltrials.gov in conjunction with an update to the protocol (September 25, 2024).
  English translated copies of the informed consent forms for both patient and physiotherapist participants are available from the corresponding author on request.
  Individual patient data (IPD) will be first made available after conclusion of data collection and publication of the study results- expected conclusion end of 2027
Access Criteria: Upon reasonable request from a credible institution or research group. Individual patient data will be shared pseudonymised upon reasonable request. This will include background data, patient reported outcome measure data and patient and physiotherapist experience measure data.

REFERENCES:
- [Background] Försäkringskassan (2023, June 20) Statistical database. Statistics related to illness. https://www.forsakringskassan.se/statistik-och-analys/statistikdatabas#!/sjuk/sjp-antal-mottagare-nettodagar-belopp
- [Background] Kallings, L. (2014). Validering av Socialstyrelsens screeningfrågor om fysisk aktivitet. The Swedish National Board of Health and Welfare. https://www.socialstyrelsen.se/globalassets/sharepoint-dokument/dokument-webb/nationella-riktlinjer/levnadsvanor-validering-av-indikatorfragor-till-patienter-om-fysisk-aktivitet.pdf
- [Background] Moseley, G. L., & Butler, D. S. (2017). Explain Pain Supercharged. NOI Group, Australia.
- [Background] Broadbent E, Wilkes C, Koschwanez H, Weinman J, Norton S, Petrie KJ. A systematic review and meta-analysis of the Brief Illness Perception Questionnaire. Psychol Health. 2015;30(11):1361-85. doi: 10.1080/08870446.2015.1070851. Epub 2015 Aug 26. PMID 26181764
- [Background] Caneiro JP, Bunzli S, O'Sullivan P. Beliefs about the body and pain: the critical role in musculoskeletal pain management. Braz J Phys Ther. 2021 Jan-Feb;25(1):17-29. doi: 10.1016/j.bjpt.2020.06.003. Epub 2020 Jun 20. PMID 32616375
- [Background] Chiarotto A, Vanti C, Cedraschi C, Ferrari S, de Lima E Sa Resende F, Ostelo RW, Pillastrini P. Responsiveness and Minimal Important Change of the Pain Self-Efficacy Questionnaire and Short Forms in Patients With Chronic Low Back Pain. J Pain. 2016 Jun;17(6):707-18. doi: 10.1016/j.jpain.2016.02.012. Epub 2016 Mar 11. PMID 26975193
- [Background] Deyo RA, Diehl AK, Rosenthal M. Reducing roentgenography use. Can patient expectations be altered? Arch Intern Med. 1987 Jan;147(1):141-5. doi: 10.1001/archinte.147.1.141. PMID 2948466
- [Background] Dube MO, Langevin P, Roy JS. Measurement properties of the Pain Self-Efficacy Questionnaire in populations with musculoskeletal disorders: a systematic review. Pain Rep. 2021 Dec 21;6(4):e972. doi: 10.1097/PR9.0000000000000972. eCollection 2021 Nov-Dec. PMID 34963996
- [Background] Emilsson M, Berndtsson I, Gustafsson PA, Horne R, Marteinsdottir I. Reliability and validation of Swedish translation of Beliefs about Medication Specific (BMQ-Specific) and Brief Illness Perception Questionnaire (B-IPQ) for use in adolescents with attention-deficit hyperactivity disorder. Nord J Psychiatry. 2020 Feb;74(2):89-95. doi: 10.1080/08039488.2019.1674376. Epub 2019 Oct 9. PMID 31596161
- [Background] Finucane LM, Downie A, Mercer C, Greenhalgh SM, Boissonnault WG, Pool-Goudzwaard AL, Beneciuk JM, Leech RL, Selfe J. International Framework for Red Flags for Potential Serious Spinal Pathologies. J Orthop Sports Phys Ther. 2020 Jul;50(7):350-372. doi: 10.2519/jospt.2020.9971. Epub 2020 May 21. PMID 32438853
- [Background] Jensen MP, Turner JA, Romano JM, Fisher LD. Comparative reliability and validity of chronic pain intensity measures. Pain. 1999 Nov;83(2):157-62. doi: 10.1016/s0304-3959(99)00101-3. PMID 10534586
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Leventhal H, Phillips LA, Burns E. The Common-Sense Model of Self-Regulation (CSM): a dynamic framework for understanding illness self-management. J Behav Med. 2016 Dec;39(6):935-946. doi: 10.1007/s10865-016-9782-2. Epub 2016 Aug 11. PMID 27515801
- [Background] Linton SJ, Nicholas M, MacDonald S. Development of a short form of the Orebro Musculoskeletal Pain Screening Questionnaire. Spine (Phila Pa 1976). 2011 Oct 15;36(22):1891-5. doi: 10.1097/BRS.0b013e3181f8f775. PMID 21192286
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Nicholas MK, McGuire BE, Asghari A. A 2-item short form of the Pain Self-efficacy Questionnaire: development and psychometric evaluation of PSEQ-2. J Pain. 2015 Feb;16(2):153-63. doi: 10.1016/j.jpain.2014.11.002. Epub 2014 Nov 14. PMID 25463701
- [Background] Olsen MF, Bjerre E, Hansen MD, Hilden J, Landler NE, Tendal B, Hrobjartsson A. Pain relief that matters to patients: systematic review of empirical studies assessing the minimum clinically important difference in acute pain. BMC Med. 2017 Feb 20;15(1):35. doi: 10.1186/s12916-016-0775-3. PMID 28215182
- [Background] Olsen MF, Bjerre E, Hansen MD, Tendal B, Hilden J, Hrobjartsson A. Minimum clinically important differences in chronic pain vary considerably by baseline pain and methodological factors: systematic review of empirical studies. J Clin Epidemiol. 2018 Sep;101:87-106.e2. doi: 10.1016/j.jclinepi.2018.05.007. Epub 2018 May 21. PMID 29793007
- [Background] Ostelo RW, Deyo RA, Stratford P, Waddell G, Croft P, Von Korff M, Bouter LM, de Vet HC. Interpreting change scores for pain and functional status in low back pain: towards international consensus regarding minimal important change. Spine (Phila Pa 1976). 2008 Jan 1;33(1):90-4. doi: 10.1097/BRS.0b013e31815e3a10. PMID 18165753
- [Background] Setchell J, Costa N, Ferreira M, Makovey J, Nielsen M, Hodges PW. Individuals' explanations for their persistent or recurrent low back pain: a cross-sectional survey. BMC Musculoskelet Disord. 2017 Nov 17;18(1):466. doi: 10.1186/s12891-017-1831-7. PMID 29149847
- [Background] Sox HC Jr, Margulies I, Sox CH. Psychologically mediated effects of diagnostic tests. Ann Intern Med. 1981 Dec;95(6):680-5. doi: 10.7326/0003-4819-95-6-680. PMID 7305144
- [Background] Vowles KE, McCracken LM, Sowden G, Ashworth J. Psychological flexibility in coping with chronic pain: further examination of the brief pain coping inventory-2. Clin J Pain. 2014 Apr;30(4):324-30. doi: 10.1097/AJP.0b013e31829ea187. PMID 23887338
- [Background] Nationella patientenkäten, Sverige Landsting och Regioner i Samverkan (2015). Rapport Analysuppdrag: Modellutveckling, utvärdering samt tidigare studier och enkäter. https://skr.se/download/18.40c889381840e60521aa1a14/1668006119029/Rapport%20Analysuppdrag_Modellutveckling,%20utv%C3%A4rdering%20samt%20tidigare%20studier%20och%20enk%C3%A4ter_2015.pdf
- [Background] Barkman, S. (2022). What do primary care professionals who meet patients with musculoskeletal pain need to facilitate the healthcare encounter? A qualitative interview study that explores the needs of professionals in primary care for knowledge and communication about pain. [Bachelor of Science (BSc) thesis. Linköping University].
- [Background] Stjärnskog, A. (2022). My pain, my needs. A qualitative interview study to investigate how primary care patients with acute and subacute musculoskeletal pain reason about their pain and what further knowledge they require. [Bachelor of Science (BSc) thesis. Linköping University].
- [Background] Öhman, S. (2022). Design guidelines for a digital educational material for patients with benign acute and sub-acute musculoskeletal pain. [Bachelor of Science (BSc) thesis. Linköping University].
- [Derived] Thompson R, Fors M, Kammerlind AS, Tingstrom P, Abbott A, Johansson K. The PainSMART project: Protocol for a research program on effectiveness, mechanisms of effect and patient-practitioner experiences of the PainSMART-strategy as an adjunct to usual primary care physiotherapy management for musculoskeletal pain. PLoS One. 2025 Jan 30;20(1):e0316806. doi: 10.1371/journal.pone.0316806. eCollection 2025. PMID 39883724

DOCUMENTS (2):
  • Study Protocol (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT06187428/Prot_002.pdf
  • Statistical Analysis Plan (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT06187428/SAP_003.pdf